CLINICAL TRIAL: NCT06934668
Title: Effect of Extracorporeal Shock Wave Therapy on Trapezius Muscle Stiffness Assessed Using Shear-Wave Elastography
Brief Title: Effect of Extracorporeal Shock Wave Therapy on Trapezius Muscle Stiffness
Acronym: ESWT-Trapezius
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Žiga Kozinc, PhD, Assistant professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWT_Trapezius
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Muscle Stiffness
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an ESWT intervention group or a control group for comparison of changes in muscle stiffness.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT (Experimental): Participants in this arm will receive a single session of extracorporeal shock wave therapy (ESWT) applied to the upper trapezius muscle (2300 waves in total).
  Interventions: Device: Extracorporeal Shock Wave Therapy
- Control group (No Intervention): Participants in this arm will not receive any therapeutic intervention. Muscle stiffness of the upper trapezius will be measured at the same time points as in the experimental group using shear-wave elastography, to evaluate the natural variability in stiffness and to serve as a comparison for the effects of ESWT.

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — A single session of focused extracorporeal shock wave therapy (ESWT) applied to the upper trapezius muscle (2300 shocks). The treatment is applied to the muscle belly region with coupling gel, without local anesthesia. The protocol is designed to assess the acute effects of ESWT on muscle stiffness measured using shear-wave elastography.
  Arms: ESWT

SUMMARY:
This study will examine whether extracorporeal shock wave therapy (ESWT) can reduce stiffness in the upper trapezius muscle. Muscle stiffness will be measured using a special ultrasound technique called shear-wave elastography (SWE), which allows researchers to assess changes in muscle properties. The aim of the study is to better understand if ESWT is effective in improving muscle function and reducing discomfort in this region. Healthy volunteers will be enrolled, and measurements will be taken before and after the ESWT treatment.

DETAILED DESCRIPTION:
This interventional study investigates the acute effects of extracorporeal shock wave therapy (ESWT) on the mechanical properties of the upper trapezius muscle, with a specific focus on muscle stiffness. Stiffness will be quantified using shear-wave elastography (SWE), a non-invasive ultrasound-based imaging modality that allows for real-time assessment of tissue elasticity.

Participants will undergo baseline SWE measurements of the upper trapezius muscle, followed by the application of a standardized ESWT protocol. Post-treatment measurements will be conducted immediately after the intervention to evaluate acute changes in stiffness. The primary objective is to determine whether a single session of ESWT induces measurable changes in muscle mechanical properties.

This study will contribute to the growing body of evidence regarding the physiological effects of ESWT on skeletal muscle tissue and its potential application in clinical and sports settings. Data collected will also support the development of future longitudinal studies assessing the therapeutic relevance of ESWT for myofascial dysfunction and musculoskeletal pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Healthy individuals with no current musculoskeletal or neurological disorders
* No history of neck or shoulder surgery
* Willingness to abstain from vigorous upper-body exercise 24 hours prior to -measurements

Exclusion Criteria:

* Presence of neck or shoulder pain within the past 3 months
* Diagnosed myofascial pain syndrome or fibromyalgia
* History of cervical spine injury or neurological conditions affecting upper limbs
* Use of analgesic or muscle relaxant medication within 48 hours prior to testing
* Pregnancy
* Contraindications to ESWT (e.g., bleeding disorders, pacemaker, malignancy in treatment area)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Trapezius Muscle Stiffness | Baseline and Immediately Post-Intervention
  Muscle stiffness of the upper trapezius will be measured using shear-wave elastography (SWE). The measure represents the shear modulus (in kilopascals) of the muscle tissue, as quantified by ultrasound imaging. Measurements will be taken with the participant in a standardized seated position, with minimal muscle activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kozinc, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No